CLINICAL TRIAL: NCT02221882
Title: A Phase 1 Study of LY3164530, a Bispecific Antibody Targeting Mesenchymal-Epithelial Transition Factor (MET) and Epidermal Growth Factor Receptor (EGFR), in Patients With Advanced or Metastatic Cancer
Brief Title: A Study of LY3164530 in Participants With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15279; I7H-MC-JNBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY3164530 (Experimental): LY3164530 in escalating dose cohorts given intravenously (IV) once on Days 1 and 15 or on Days 1, 8, 15, and 22 of a 28-day cycle. Participants may continue to receive study drug until discontinuation criteria are met.
  Interventions: Drug: LY3164530

INTERVENTIONS:
Drug: LY3164530 — Administered IV.

SUMMARY:
The main purpose of this study is to evaluate the safety of a study drug known as LY3164530 in participants with cancer that is advanced and/or has spread to another part(s) of the body.

ELIGIBILITY:
Inclusion Criteria

* Have advanced or metastatic cancer and be an appropriate candidate for experimental therapy.
* Have adequate organ function.
* Prior Treatments:

  * Systemic treatments: Must have discontinued previous systemic treatments for cancer and recovered from the acute effects of therapy. Participants must have discontinued:

    * Cytotoxic therapies or targeted agents that are small molecule inhibitors for 5 half-lives or at least 28 days.
    * Mitomycin-C or nitrosourea therapy for at least 42 days and biologic agents for at least 28 days.
  * Radiation therapy and surgery must be completed 4 weeks prior to therapy, except for limited field radiation therapy, which must be completed 2 weeks before therapy.
* If participant is of reproductive potential, must agree to use medically approved contraceptive precautions during the study and for three months following the last dose of study drug.
* If the participant is a female of childbearing potential, must have had a negative serum or urine pregnancy test within 14 days of the first dose of study drug and must not be breast feeding.

Exclusion Criteria:

* Must not have taken an unapproved drug as treatment for any indication within the last 28 days prior to starting study treatment.
* Must not have an active symptomatic fungal, bacterial or viral infection, including human immunodeficiency virus (HIV) or Hepatitis A, B, or C.
* Must not have a serious preexisting medical conditions or concomitant disorders.
* Must not have leukemia.
* Must not have QT interval of >470 millisecond.
* Must not have a serious cardiac condition, such as congestive heart failure, unstable angina pectoris, or heart attack within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-08; Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The START Center for Cancer Care, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants, who completed at least 1 cycle of treatment or discontinued due to an adverse event during Cycle 1 and completed the required post-treatment safety assessment, were considered to have completed the study.
Groups:
- 300 mg LY3164530 Schedule 1: 300 mg LY3164530 given intravenously (IV) on Days 1 and 15 of each 28 day cycle.
- 600 mg LY3164530 Schedule 1: 600 mg LY3164530 given IV on Days 1, and 15 of each 28 day cycle.
- 1000 mg LY3164530 Schedule 1: 1000 mg LY3164530 given IV on Days 1 and 15 of each 28 day cycle.
- 1250 mg LY3164530 Schedule 1: 1250 mg LY3164530 given IV on Days 1 and 15 of each 28 day cycle.
- 500 mg LY3164530 Schedule 2: 500 mg LY3164530 given IV on Days 1, 8, 15, and 22 of each 28 day cycle.
- 600 mg LY3164530 Schedule 2: 600 mg LY3164530 given IV on Days 1, 8, 15, and 22 of each 28 day cycle.
Period: Overall Study
Arm/Group | 300 mg LY3164530 Schedule 1 | 600 mg LY3164530 Schedule 1 | 1000 mg LY3164530 Schedule 1 | 1250 mg LY3164530 Schedule 1 | 500 mg LY3164530 Schedule 2 | 600 mg LY3164530 Schedule 2
Started | 3 | 3 | 11 | 3 | 5 | 4
Received at Least One Dose of Study Drug | 3 | 3 | 11 | 3 | 5 | 4
Completed | 3 | 2 | 7 | 1 | 3 | 2
Not Completed | 0 | 1 | 4 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 2 | 2 | 2
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 mg LY3164530 Schedule 1 | 600 mg LY3164530 Schedule 1 | 1000 mg LY3164530 Schedule 1 | 1250 mg LY3164530 Schedule 1 | 500 mg LY3164530 Schedule 2 | 600 mg LY3164530 Schedule 2 | Total
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 5 | 4 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5 | 2 | 3 | 2 | 17
  >=65 years | 1 | 0 | 6 | 1 | 2 | 2 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 2 | 2 | 3 | 12
  Male | 1 | 3 | 8 | 1 | 3 | 1 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 3 | 0 | 1 | 1 | 7
  Not Hispanic or Latino | 3 | 1 | 8 | 3 | 4 | 3 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 11 | 3 | 5 | 3 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 11 | 3 | 5 | 4 | 29

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose of LY3164530: Maximum Tolerated Dose (MTD)
Description: Recommended Phase 2 Dose of LY3164530: MTD
Time Frame: Cycle 1 (Cycle = 28 days)
Population: All participants who receive at least one dose of study drug.
Measure: Number; unit: milligrams (mg)
Groups:
- Schedule 1: LY3164530 in escalating dose cohorts of 300mg, 600mg, 1000mg and 1250mg given intravenously (IV) once on Days 1, 8, 15, and 22 of a 28-day cycle.
- Schedule 2: LY3164530 in escalating dose cohorts of 500 mg or 600 mg given intravenously (IV) once on Days 1 and 15 of a 28-day cycle.
Arm/Group | Schedule 1 | Schedule 2
Number analyzed (Participants) | 20 | 9
milligrams (mg) | 1000 | 500

2. Secondary Outcome: Maximum Serum Concentration (Cmax) of LY3164530 Epidermal Growth Factor Receptor (EGFR) Specific ELISA Assay
Description: Cmax in Schedule (Sched) 1 Cycle 1 (C1) and Cycle 2 (C2) and Sched. 2 C1 and C2 dose escalation based on EGFR specific ELISA assay.
  Pharmacokinetic (PK) Time Frame Schedule 1:Cycle 1 and 2 (Day 1): Predose; Mid-infusion; End of infusion; 2 hours (hrs), 4hrs, 6hrs, 24 ±4hrs post-infusion; Day 3: anytime during day; Day 8 ±1 : anytime during day. Day 15: Pre-dose, End of infusion; 2hrs, 4hrs, 6hrs post-infusion; Day 22 ±2: anytime during day. Cycles 3-6: Pre-dose, End of infusion.
  PK Time Frame: Schedule 2: Cycle 1 and 2 (Day 1): Predose; Mid-infusion; End of infusion; 2hrs, 4hrs, 6hrs, 24 ±4hrs post-infusion (Cycle 1); Day 3: anytime during day; Day 8: Pre-dose; End of infusion; Day 22: Pre-dose; End of infusion; 2hrs, 4hrs, 6hrs, 24 ±4hrs post-infusion (Cycle 1); Day 24: anytime during day. Cycles 3-6: Pre-dose; End of Infusion.
Time Frame: Cycle 1 predose (Day 1) up to Cycle 6 end of infusion (Day 1)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL )
Arm/Group | 300 mg LY3164530 Schedule 1 | 600 mg LY3164530 Schedule 1 | 1000 mg LY3164530 Schedule 1 | 1250 mg LY3164530 Schedule 1 | 500 mg LY3164530 Schedule 2 | 600 mg LY3164530 Schedule 2
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 5 | 4
microgram per milliliter (µg/mL )
  Schedule 1 Cycle 1 Day 1; Schedule 2 Cycle 1 Day 1 | 85.1 (38) | 122 (12) | 367 (52) | 496 (30) | 226 (20) | 255 (21)
  Schedule 1 Cycle 1 Day 15;Schedule 2 Cycle 1Day 22: number analyzed (Participants) | 2 | 3 | 11 | 3 | 5 | 3
  Schedule 1 Cycle 1 Day 15;Schedule 2 Cycle 1Day 22 | NA (NA) — Geometric mean and coefficient of variation (CV) not calculated for 2 participants; individual participants values reported: 119.55 and 66.36. | 147 (15) | 348 (34) | 615 (38) | 262 (35) | 350 (20)
  Schedule 1 Cycle 2 Day 1; Schedule 2 Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 9 | 1 | 5 | 2
  Schedule 1 Cycle 2 Day 1; Schedule 2 Cycle 2 Day 1 | 72.19 (NA) — Coefficient of variation was not calculated for 1 participant. | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual participants values reported: 115.02 and 135.38. | 357 (35) | 468.9 (NA) — Coefficient of variation was not calculated for 1 participant. | 270 (32) | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual participants values reported: 547.9 and 431.2.

3. Secondary Outcome: Maximum Serum Concentration (Cmax) of LY3164530 Mesenchymal-Epithelial Transition Factor (MET) Specific ELISA Assay
Description: Cmax in Schedule 1 Cycles 1 and 2 and Schedule 2 Cycles 1 and 2 based on the MET-specific ELISA assay.
  Pharmacokinetic (PK) Time Frame Schedule 1:Cycle 1 and 2 (Day 1): Predose; Mid-infusion; End of infusion; 2 hours (hrs), 4hrs, 6hrs, 24 ±4hrs post-infusion; Day 3: anytime during day; Day 8 ±1 : anytime during day. Day 15: Pre-dose, End of infusion; 2hrs, 4hrs, 6hrs post-infusion; Day 22 ±2: anytime during day. Cycles 3-6: Pre-dose, End of infusion.
  PK Time Frame: Schedule 2: Cycle 1 and 2 (Day 1): Predose; Mid-infusion; End of infusion; 2hrs, 4hrs, 6hrs, 24 ±4hrs post-infusion (Cycle 1); Day 3: anytime during day; Day 8: Pre-dose; End of infusion; Day 22: Pre-dose; End of infusion; 2hrs, 4hrs, 6hrs, 24 ±4hrs post-infusion (Cycle 1); Day 24: anytime during day. Cycles 3-6: Pre-dose; End of Infusion.
Time Frame: Cycle 1 predose (Day 1) up to Cycle 6 end of infusion (Day 1)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | 300 mg LY3164530 Schedule 1 | 600 mg LY3164530 Schedule 1 | 1000 mg LY3164530 Schedule 1 | 1250 mg LY3164530 Schedule 1 | 500 mg LY3164530 Schedule 2 | 600 mg LY3164530 Schedule 2
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 5 | 4
µg/mL
  Schedule 1 Cycle 1 Day 1; Schedule 2 Cycle 1 Day 1 | 82.5 (41) | 124 (15) | 365 (46) | 498 (33) | 208 (23) | 221 (21)
  Schedule 1 Cycle 1 Day 15;Schedule 2 Cycle 1Day 22: number analyzed (Participants) | 2 | 3 | 11 | 3 | 5 | 3
  Schedule 1 Cycle 1 Day 15;Schedule 2 Cycle 1Day 22 | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual values reported: 127.21 and 73.21. | 136 (12) | 346 (33) | 587 (35) | 260 (32) | 317 (17)
  Schedule 1 Cycle 2 Day 1; Schedule 2 Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 9 | 1 | 5 | 2
  Schedule 1 Cycle 2 Day 1; Schedule 2 Cycle 2 Day 1 | 72.32 (NA) — The coefficient of variation was not calculated for 1 participant. | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual participants values reported:123.84 and 143.68. | 353 (27) | 400.9 (NA) — The coefficient of variation was not calculated for 1 participant. | 258 (27) | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual participants values reported: 541.5 and 347.0.

4. Secondary Outcome: Area Under the Serum Concentration-Time Curve (AUC[0-τ]) of LY3164530 EGFR Specific ELISA Assay
Description: Area under the serum concentration-time curve of LY3164530 over the dosing interval (AUC[0-τ]) from time 0 to 336 hours (τ) [Schedule 1] or from time 0-168 hours (τ) [Schedule 2].
  Pharmacokinetic (PK) Time Frame Schedule 1:Cycle 1 and 2 (Day 1): Predose; Mid-infusion; End of infusion; 2 hours (hrs), 4hrs, 6hrs, 24 ±4hrs post-infusion; Day 3: anytime during day; Day 8 ±1 : anytime during day. Day 15: Pre-dose, End of infusion; 2hrs, 4hrs, 6hrs post-infusion; Day 22 ±2: anytime during day. Cycles 3-6: Pre-dose, End of infusion.
  PK Time Frame: Schedule 2: Cycle 1 and 2 (Day 1): Predose; Mid-infusion; End of infusion; 2hrs, 4hrs, 6hrs, 24 ±4hrs post-infusion (Cycle 1); Day 3: anytime during day; Day 8: Pre-dose; End of infusion; Day 22: Pre-dose; End of infusion; 2hrs, 4hrs, 6hrs, 24 ±4hrs post-infusion (Cycle 1); Day 24: anytime during day. Cycles 3-6: Pre-dose; End of Infusion.
Time Frame: Cycle 1 predose (Day 1) up to Cycle 6 end of infusion (Day 1)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*milliliter per hour(µg*mL/hr)
Arm/Group | 300 mg LY3164530 Schedule 1 | 600 mg LY3164530 Schedule 1 | 1000 mg LY3164530 Schedule 1 | 1250 mg LY3164530 Schedule 1 | 500 mg LY3164530 Schedule 2 | 600 mg LY3164530 Schedule 2
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 5 | 4
micrograms*milliliter per hour(µg*mL/hr)
  Schedule 1 Cycle 1 Day 1; Schedule 2 Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 11 | 3 | 4 | 4
  Schedule 1 Cycle 1 Day 1; Schedule 2 Cycle 1 Day 1 | 5580 (28) | 9870 (23) | 37000 (42) | 57500 (28) | 16700 (37) | 19800 (21)
  Schedule 1 Cycle 1 Day 15;Schedule 2 Cycle 1 Day 2: number analyzed (Participants) | 2 | 3 | 10 | 3 | 5 | 3
  Schedule 1 Cycle 1 Day 15;Schedule 2 Cycle 1 Day 2 | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual values reported: 13100 and 7170. | 13700 (15) | 42700 (39) | 81400 (31) | 25500 (35) | 34900 (31)
  Schedule 1 Cycle 2 Day 1; Schedule 2 Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 8 | 1 | 5 | 2
  Schedule 1 Cycle 2 Day 1; Schedule 2 Cycle 2 Day 1 | 6690 (NA) — The coefficient of variation was not calculated for 1 participant. | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual values reported: 12100 and 13300. | 43000 (55) | 51500 (NA) — The coefficient of variation was not calculated for 1 participant. | 26300 (35) | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual values reported: 31900 and 41300.

5. Secondary Outcome: Area Under the Serum Concentration-Time Curve (AUC[0-τ]) of LY3164530 MET Specific ELISA Assay
Description: as for outcome 4
Time Frame: Cycle 1 predose (Day 1) up to Cycle 6 end of infusion (Day 1)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | 300 mg LY3164530 Schedule 1 | 600 mg LY3164530 Schedule 1 | 1000 mg LY3164530 Schedule 1 | 1250 mg LY3164530 Schedule 1 | 500 mg LY3164530 Schedule 2 | 600 mg LY3164530 Schedule 2
Number analyzed (Participants) | 3 | 3 | 11 | 3 | 5 | 4
µg*hr/mL
  Schedule 1 Cycle 1 Day 1; Schedule 2 Cycle 1 Day 1 | 6150 (26) | 10900 (27) | 37500 (41) | 57300 (31) | 16300 (22) | 17500 (20)
  Schedule 1 Cycle 1 Day 15;Schedule 2 Cycle 1 Day 2: number analyzed (Participants) | 2 | 3 | 11 | 3 | 5 | 3
  Schedule 1 Cycle 1 Day 15;Schedule 2 Cycle 1 Day 2 | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual values reported: 12200 and 7260. | 12900 (14) | 43000 (34) | 82000 (33) | 24800 (29) | 31200 (30)
  Schedule 1 Cycle 2 Day 1; Schedule 2 Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 8 | 1 | 5 | 2
  Schedule 1 Cycle 2 Day 1; Schedule 2 Cycle 2 Day 1 | 6800 (NA) — The coefficient of variation was not calculated for 1 participant. | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual values reported: 11800 and 13300. | 44700 (45) | 46400 (NA) — The coefficient of variation was not calculated for 1 participant. | 24800 (34) | NA (NA) — Geometric mean and CV not calculated for 2 participants; individual values reported: 29500 and 36700.

6. Secondary Outcome: Number of Participants With Tumor Response
Description: Number of Participants with Tumor Response
Time Frame: Baseline Through Study Completion (Up to 6 Months)
Population: All participants who received at least one dose of study drug and had at least one post-baseline tumor assessment.
Measure: Count of Participants; unit: Participants
Groups:
- 300mg LY3164530 Schedule 1: 300 mg LY3164530 given intravenously (IV) on Days 1 and 15 of each 28 day cycle.
- 1250 mg LY3164530 Schedule 1: 1000 mg LY3164530 given IV on Days 1 and 15 of each 28 day cycle.
Arm/Group | 300mg LY3164530 Schedule 1 | 600 mg LY3164530 Schedule 1 | 1000 mg LY3164530 Schedule 1 | 1250 mg LY3164530 Schedule 1 | 500 mg LY3164530 Schedule 2 | 600 mg LY3164530 Schedule 2
Number analyzed (Participants) | 3 | 3 | 9 | 3 | 5 | 4
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 2 | 1
  Stable Disease | 1 | 1 | 6 | 1 | 1 | 2
  Progressive Disease | 2 | 2 | 3 | 2 | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline Through Study Completion (Up to 6 Months)
Arm/Group | 300 mg LY3164530 Schedule 1 | 600 mg LY3164530 Schedule 1 | 1000 mg LY3164530 Schedule 1 | 1250 mg LY3164530 Schedule 1 | 500 mg LY3164530 Schedule 2 | 600 mg LY3164530 Schedule 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 0/11 | 0/3 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 3/11 | 0/3 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 11/11 | 3/3 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg LY3164530 Schedule 1 (N=3) | 600 mg LY3164530 Schedule 1 (N=3) | 1000 mg LY3164530 Schedule 1 (N=11) | 1250 mg LY3164530 Schedule 1 (N=3) | 500 mg LY3164530 Schedule 2 (N=5) | 600 mg LY3164530 Schedule 2 (N=4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg LY3164530 Schedule 1 (N=3) | 600 mg LY3164530 Schedule 1 (N=3) | 1000 mg LY3164530 Schedule 1 (N=11) | 1250 mg LY3164530 Schedule 1 (N=3) | 500 mg LY3164530 Schedule 2 (N=5) | 600 mg LY3164530 Schedule 2 (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (3) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trichomegaly (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (9)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (2)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral contusion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 2 (3)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue eruption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 3 (5) | 2 (3) | 3 (7) | 2 (15)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (4) | 0 (0) | 4 (5) | 0 (0) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 2 (4) | 2 (2)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (5) | 1 (1) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 1 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (10) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (8) | 1 (2) | 3 (11) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (26) | 2 (7) | 5 (17) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Horner's syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 1 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal mucosal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (7) | 1 (1) | 1 (2) | 1 (4) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 9 (27) | 1 (2) | 4 (15) | 3 (13)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 4 (7) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-09-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT02221882/Prot_000.pdf
  • Statistical Analysis Plan (2014-06-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT02221882/SAP_001.pdf